CLINICAL TRIAL: NCT04135729
Title: Body Image and Mental Health Symptoms in Personal Trainers and Group Instructors
Brief Title: Mental Health in Fitness Instructors
Status: Completed | Type: Observational
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: Ostfold University College (Other); University College of Southeast Norway (Other)
Responsible Party: Principal Investigator, Professor Jorunn Sundgot-Borgen, Professor, Norwegian School of Sport Sciences
Other Study IDs: 19/00742; 28855 (Other: Regional Committees for Medical and Health Research Ethics)
Record Dates: First submitted 2019-10-20; First posted 2019-10-23 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Mental Health Wellness 1; Depression, Anxiety; Eating Disorders; Eating Behavior; Body Image; Sexual Harassment; Exercise Addiction; Weight Change, Body; Weight Loss; Weight Gain; Leanness; Amenorrhea; Dietary Habits; Body Image Disturbance; Thinness
Keywords: Mental health; Eating disorders; Depression; Anxiety; Body dissatisfaction; Body image; Thinness; Leanness; Muscularity; Compulsive exercise; Eating behavior; Dieting; Exercise; Sexual harassment
MeSH Terms: conditions — Depression; Anxiety Disorders; Feeding and Eating Disorders; Feeding Behavior; Sexual Harassment; Body Weight Changes; Weight Loss; Weight Gain; Thinness; Amenorrhea; Psychological Well-Being; Compulsive Exercise; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Personal trainer (PT): Cross-sectional study on mental health symptoms in personal trainers
- Group instructors (GI): Cross-sectional study on mental health symptoms in group instructors
- Combined instructors (PT + GI): Cross-sectional study on mental health symptoms in personal trainers

SUMMARY:
The aim of this project is to improve the evidence-base regarding lifestyle and mental health symptoms among fitness instructors. A national cohort of fitness instructors will be invited to participate in this study by responding to an online questionnaire. The questionnaire will consist of items regarding exercise, nutrition, eating disorders, the menstrual cycle, depression, anxiety, body dissatisfaction and satisfaction, drive for muscularity and leanness, and experiences of sexual harassment. Findings from this study will provide an evidence-base for initiatives to improve/optimize mental health among fitness instructors, and also in the process of developing fitness centres to a core partner in public health and health promotion work.

DETAILED DESCRIPTION:
Previous research has shown that prevalence of self-reported eating disorders vary from 5-40% among group fitness instructors. Most of these studies were conducted more than 10 years ago, hence the potential impact of social media on the fitness instructors' body image and mental health symptoms has therefore not been taken into account. Recent studies reveal that social media is a significant contributor for perceived body image and for eating and exercise-related disturbances. A more recent Norwegian study from 2015 found a prevalence of self-reported eating disorders of 4.8% and 4.3% among female and male group fitness instructors, respectively. However, major limitations with this previous study was the low sample size (n=107), few men included, not being national representative (i.e. only recruiting from a smaller geographical area), and the lack of instruments assessing body awareness of muscularity and leanness instead of thinness.

The fitness industry has great potential as a public health collaborator, and to improve physical activity level and public health status. However, this potential can be flawed by instructors complying with a culture idealizing unhealthy attitudes, motivation and behaviour with regards to nutrition, exercise and body image. This is a culture also potentially being underlined by the new exercise concepts and titles brought forward by the fitness industry, emphasizing body ideals and appearance, and body weight control. An additional concern to the mental health of fitness instructors, are the increase in reports of sexual harassment.

The high prevalence of perceived negative body image and disordered eating among fitness instructors, reports of sexual harassment, and the focus on appearance and control of body shape in the fitness industry, causes concern for the mental health of the employees (i.e. fitness instructors). Hence, this cohort study aims to map the prevalence of mental health symptoms in a national cohort of fitness instructors.

ELIGIBILITY:
Inclusion Criteria:

* Operating as a fitness instructor (personal trainer or group instructor) during autumn 2019
* Age above 18 years
* Living and operating in Norway
* Understanding and communicating with Norwegian language

Exclusion Criteria:

* Not engaged as a fitness instructor at recruitment time (autumn 2019)
* Age below 18 years of age
* Not living and/or operating in Norway
* Only speaking/communicating in foreign language (i.e. not Norwegian language)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All operating fitness instructors working at fitness facilities/gym's in Norway during autumn 2019 are recruited by information in social media, by information given directly to CEO/administration of facilities listed by the cooperative in Norway, Virke Trening, and by information given directly to gym facilities identified by other means in Norway.
Sampling Method: Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Body image | Autumn 2019
  Body image in fitness instructors (personal trainers and group instructors) by Body Appreciation Scale-2 (BAS-2). The scale comprises 10 items rated on a 5-point scale, ranging from 1 (Never) to 5 (Always), with higher total scoring indicating more positive body appreciation.
Eating disorders | Autumn 2019
  Prevalence of eating disorders in fitness instructors (personal trainers and group instructors) by Eating disorders Examination questionnaire (EDE-q). The questionnaire has 6 items with open scorings reporting frequency of symptoms, and 22 items scored on a likert scale from 0-6 (no days - all days). The questionnaire has a total score and four subscales, with higher scorings (ranging from 0-6) indicative of higher severity.

SECONDARY OUTCOMES:
Depression | Autumn 2019
  Symptoms of depression in fitness instructors (personal trainers and group instructors) by Beck Depression Inventory (BDI-1a). It consists of 21 items scored on a 4-point Likert scale ranging from 0 (not at all) to 3 (extreme). Total score range is 0-63, and a cutoff score of ≥21 is recommended for use to detect a clinically significant episode of major depression.
Mental health symptoms | Autumn 2019
  Symptoms of mental health symptoms in fitness instructors (personal trainers and group instructors) by Symptom Check List (SCL-10). The 10-item questionnaire measures symptoms of anxiety and depression with a likert scale ranging from 0-4 (not at all - very much), with higher scoring meaning higher clinical severity.
Drive for leanness | Autumn 2019
  Symptoms of drive for leanness in fitness instructors (personal trainers and group instructors) by Drive for Leanness scale. It constitutes 6 questions scored by a 6 point scale ranging from never (1) to always (6) with a possible total score 0-36, and in which higher score is indicative of greater investment in leanness.
Drive for muscularity | Autumn 2019
  Symptoms of drive for muscularity in fitness instructors (personal trainers and group instructors) by Drive for Muscularity Scale. It constitutes seven questions scored on a 6 points scale ranging from (1) always to (6) never, uses a reversed coding in analysis, and has a total score of 15-90 (high score means higher DM).
Compulsive Exercise | Autumn 2019
  Symptoms of compulsive exercise in fitness instructors (personal trainers and group instructors) by Compulsive exercise test (CET). CET is a 24-item instrument scored on a 5-point Likert scale (0 = never true, 5 = always true), and evaluated with five different subscale mean scores (avoidance and rule driven behaviour, weight control exercise, mood improvement, lack of exercise enjoyment, and exercise rigidity), and a global score summing the means of subscales (score range 0-30).
Drive for thinness | Autumn 2019
  Symptoms of drive for thinness in fitness instructors (personal trainers and group instructors) by Drive for Thinness subscale (DT) of Eating Disorder Inventory (EDI-3). The subscales constitutes 7 of the totally 91 questions in the EDI-3, and is scored on a likert scale from 0-4, with higher scoring meaning higher clinical severity, and a suggested clinical cutoff of 14.
Sexual harassment | Autumn 2019
  Experience of sexual harassment in professional work by fitness instructors (personal trainers and group instructors). This is screened by questions on experiences of harassment of different character (comments, characteristic bodily movements, or physical touch or abuse), and scored on a scale by alternatives; never, yes-by collegues, yes-by clients, yes-by leaders.
Sociocultural Attitudes Towards Appearance Questionnaire | Autumn 2019
  Sociocultural Attitudes Towards Appearance in fitness instructors (personal trainers and group instructors). The questionnaire has subscales that assess internalization (general, athlete), pressures, and information, and is scored from 1-5 (def. disagree - def. agree), with higher scorings indicating higher clinical severity.
Eating behavior | Autumn 2019
  Symptoms of eating behavior in fitness instructors (personal trainers and group instructors) by Three Factor Eating Questionnaire (TFE-q 21). TFE-q measures symptoms of cognitive restrictive eating (RE, 6 items), emotional eating (EE, 6 items), and uncontrolled eating (UE, 9 items). It constitutes 20 questions rating agreements to different assertions by score of 1-4, and one question rating agreement by 1-8 points. The total subscale scores may be presented as raw scores, or as transformed scores (scale 0-100), and higher scorings means higher clinical severity.

OTHER OUTCOMES:
Body weight history | Autumn 2019
  Body weight history (i.e. body weight fluctuations) in fitness instructors, reported by selfreported minimum and maximum adult bodyweight.
Dieting behavior | Autumn 2019
  Dieting behavior: questions on whether they aim to reduce og gain body weight, and by which methods (several choices), by what guidance (several choices), what frequency of meal intake per day, and whether they use supplements (and if so: which supplements).
Diagnosis of eating disorder | Autumn 2019
  selfreported history of eating disorders by fitness instructors
Experiences of body image idealization | Autumn 2019
  Personal experiences of body image idealization in professional career by fitness instructors. Do they experience body image idealization (yes/no), in what areas of professional work (by clients, by colleagues, by the work facility culture), does it affect them positively or negatively, do they recognize any preventive or awarness-raising work from the administration/workplace, is this procedure actually complied with.
Social Media | Autumn 2019
  Use of, and experienced influence by, social media in fitness instructors. Selfreported use of social media (which social media), their motivation in doing so, and for what purposes/motivations social media is followed by oneself.

CONTACTS AND LOCATIONS:
Overall Officials: Jorunn Sundgot-Borgen, PhD, Principal Investigator — Norwegian School of Sport Sciences
Locations (1):
- Norwegian school of sport sciences, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Data is held within the group of scientists, but sharing may be evaluated on request.